CLINICAL TRIAL: NCT07228182
Title: Effect of High-Intensity Transcranial Alternating Current Stimulation on Gambling Disorder: A Randomized Controlled Trial
Acronym: HITACSRCT-GD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDu-017
Record Dates: First submitted 2025-11-10; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gambling Disorder
Keywords: High-Intensity Transcranial Alternating Current Stimulation, Gambling disorder.
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention group for gambling addiction (Experimental): A 40-minute transcranial alternating current stimulus intervention of real stimulus is conducted twice a day (at least 3 hours apart) for a total of 10 days in the intervention group of gambling addiction.
  Interventions: Device: HI-tACS
- Sham stimulation (Sham Comparator): A 40-minute transcranial alternating current stimulus intervention of sham stimulus is conducted twice a day (at least 3 hours apart) for a total of 10 days in the intervention group of gambling addiction.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: HI-tACS — Three conductive electrodes are placed overhead. In the 10/20 international placement system, a 4.45 9.53 cm electrode is placed on the forehead corresponding to Fpz, Fp1 and Fp2. Two 3.18 3.81 cm electrodes are placed on the mastoid region of each side. The tACS stimulation waveform includes ramp-up and ramp-down periods of 180 and 12 s, respectively. The frequency of stimulation is 77.5Hz, and the current is 15mA.
  Arms: Intervention group for gambling addiction
Device: Sham stimulation — Three conductive electrodes are placed overhead. In the 10/20 international placement system, a 4.45 9.53 cm electrode is placed on the forehead corresponding to Fpz, Fp1 and Fp2. Two 3.18 3.81 cm electrodes are placed on the mastoid region of each side. The appearance of the above-mentioned equipment is identical to that of the real stimulation group devices, but it only simulates the electrical sensation produced at the beginning and end of stimulation.
  Arms: Sham stimulation

SUMMARY:
The investigators assume that transcranial Alternating Current Stimulation (tACS) could improve gambling disorder patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. This study intends to validate the effect of tACS treatment, which has been discovered in the previous pilot study. Three-month follow-up assessment will be conducted to test the changing of the executive-control function and its mechanism.

DETAILED DESCRIPTION:
Gambling disorder is become a major social and public health problem in China. Executive-control dysfunction is the main symptom of behavioral addiction like gambling disorder. Previous studies have demonstrated the relationship between cognitive dysfunction and prefrontal-ventral striatum pathway. Studies have shown that abnormal phase synchronization and phase-amplitude coupling (PAC) induced the impairment of cognition, and transcranial Alternating Current Stimulation (tACS) could improve executive-control function by adjusting the abnormal synchronization. However, it has not been verified among gambling disorder patients. The investigators assume that tACS could improve gambling disorder patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. This study intends to test the effect of tACS treatment, which has been discovered in the previous pilot study. Three-month follow-up assessment will be conducted to test the changing of the executive-control function and its mechanism. This study will provide a practical and theoretical basis for developing a novel treatment for gambling disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60, male or female, with 9 or more years of education, and able to complete questionnaire evaluation and behavioral tests;
* Meet DSM-5 (Diagnostic and Statistical Manual of mental disorders，DSM) diagnostic criteria for gambling disorder;
* Have gambled for at least one year (at least once a week);
* Normal vision and hearing, or within the normal range after correction;
* Agree to cooperate in the follow-up evaluation;
* No metal implantation in the head, no history of nerve problems or head injury, and no skin sensitivity.

Exclusion Criteria:

* Have severe cognitive impairment, such as a history of head trauma, -cerebrovascular disease, epilepsy, etc.;
* Have used drugs promoting cognitive function in the last 6 months;
* Have impaired intelligence (Intelligence Quotient<70);
* Abuse or dependence of psychoactive substances (except nicotine) in the last 5 years.

Ages: 16 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Change of the gambling symptoms | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Gambling symptom severity will be measured by the Pathological Gambling Yale-Brown Obsessive Compulsive Scale (PG-YBOCS). The total score of PG-YBOCS ranges from 0 to 40, in which higher scores indicate more severe pathological gambling symptoms.

SECONDARY OUTCOMES:
Change of depressive symptoms | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Depressive symptoms will be measured by the 17-item Hamilton Depression Rating Scale (HAMD-17). The total score of HAMD-17 ranges from 0 to 52, in which higher scores mean a higher severity of depressive symptoms.
Change of anxiety symptoms | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Anxiety symptoms will be measured by the 14-item Hamilton Anxiety Rating Scale (HAMA-14). The total score of HAMA-14 ranges from 0 to 56, in which higher scores mean a higher severity of anxiety symptoms.
Change of the sleep quality | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). The total score of PSQI ranges from 0 to 21, in which higher scores mean poorer sleep quality.
Change of the gambling craving | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Gambling craving will be measured by the gambling craving Visual Analog Scale (VAS). The total score of VAS ranges from 0 to 10, in which higher scores mean a higher level of gambling craving.
Side effect of the modulation | Immediately after the intervention
  Side effects will be measured by the Treatment Emergent Symptom Scale (TESS). The total score of TESS varies depending on symptom severity, in which higher scores indicate more significant adverse reactions.
Change of the self-control ability | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Self-control ability will be measured by the Self-Control Scale (SCS). Higher scores of SCS indicate better self-regulation and impulse control.
Change of the gambling symptom severity | Baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Gambling symptom severity will be measured by the Gambling Symptom Assessment Scale (G-SAS). The total score of G-SAS ranges from 0 to 48, in which higher scores mean more severe gambling-related symptoms.
Change of the risky decision-making performance | Baseline, two weeks after the intervention.
  Risky decision-making performance will be assessed using the Balloon Analogue Risk Task (BART). Higher average pumps in the BART indicate greater risk-taking propensity. Feedback-related negativity (FRN) will be recorded using electroencephalography (EEG), with larger amplitude typically reflecting enhanced sensitivity to negative feedback.
  Pig dice game will be administered during functional magnetic resonance imaging (fMRI) scanning to assess risk-taking decision-making. Higher frequency of continued dice rolls indicates greater risk propensity. Neural activity in the prefrontal cortex and striatum will be analyzed, with increased activation typically associated with risk evaluation and reward processing.
Change of the inhibitory control performance | Baseline, two weeks after the intervention.
  Stop-signal task (SST) will be employed to measure inhibitory control. Longer stop-signal reaction times (SSRT) indicate poorer response inhibition. The N2/P3 components will be recorded using electroencephalography (EEG), with enhanced N2 amplitude and reduced P3 amplitude typically reflecting greater cognitive conflict and inhibitory processing efficiency, respectively.
Change of the resting state neural activity. | Baseline, two weeks after the intervention.
  Resting-state functional magnetic resonance imaging (rsfMRI) will be used to assess intrinsic brain connectivity. Lower amplitude of low-frequency fluctuations (ALFF) and reduced functional connectivity (FC) within the default mode network (DMN) may reflect altered neural efficiency. Resting-state electroencephalography (rsEEG) will be employed to measure spontaneous neural oscillations. Enhanced theta/beta ratio and reduced alpha power may indicate compromised regulatory control and cortical arousal, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No